CLINICAL TRIAL: NCT04545164
Title: Computer Aided Screening for Tuberculosis in Low Resource Environments
Acronym: CASTLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Liverpool School of Tropical Medicine (Other); Kamuzu University of Health Sciences (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17799
Record Dates: First submitted 2020-09-01; First posted 2020-09-10 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-05

CONDITIONS: Tuberculosis Infection; HIV Infections
MeSH Terms: conditions — Latent Tuberculosis; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Participants in the usual care arm will receive no specific trial intervention. Usual care includes tests routinely available at Zomba Central Hospital, including (but not limited to) conventional (plain film) chest X-ray, urine Alere LAM and sputum Xpert Mtb/Rif on treating clinician request.
- DCXR-CAD and FujiLAM and usual care (Experimental): Participants randomized to the intervention arm will receive TB screening using DCXR-CAD and urine FujiLAM. The CAD score and FujLAM results will be appended into their medical notes for treating clinicians to see. If patients have a CAD score above a pre-determined threshold the study team will attempt to collect sputum for Xpert Mtb/Rif. Chest X-ray images will be available for clinicians to view. This is in addition to usual care (detailed above).
  Interventions: Diagnostic Test: CAD4TB; Diagnostic Test: FujiLAM
- Diagnostic cohort (Other): Patients in the observational enhanced diagnostic arm will receive an enhanced package of diagnostics. This is a smaller arm (1 in 9 of all clusters) and is observational only - participants in this arm do not contribute to trial outcomes.
  Interventions: Diagnostic Test: CAD4TB; Diagnostic Test: FujiLAM

INTERVENTIONS:
Diagnostic Test: CAD4TB — CAD4TB is a Computer Aided Diagnosis (CAD) image processing algorithm that can aid interpretation of Chest X-ray images to accurately detect tuberculosis.
  Arms: DCXR-CAD and FujiLAM and usual care; Diagnostic cohort
Diagnostic Test: FujiLAM — Fujifilm SILVAMP TB LAM is a high sensitivity test for mycobacterial lipoarabinomannan (LAM) in urine samples.
  Arms: DCXR-CAD and FujiLAM and usual care; Diagnostic cohort

SUMMARY:
People living with HIV (PLHIV) who require admission to hospital in WHO Africa region have poor outcomes. TB is very common in this group, but can be difficult to diagnose.

The CASTLE trial aims to determine whether systematic screening for tuberculosis using digital chest X-ray with computer-aided diagnosis (DCXR-CAD) plus urine lipoarabinomannan testing with Fujifilm SILVAMP TB LAM (FujiLAM) plus usual care can improve admission outcomes for hospitalised PLHIV, compared to usual care alone.

Our study is a single centre, unblinded, cluster-randomised (by day of admission) trial of DCXR-CAD plus FujiLAM plus usual care vs. usual care alone for screening for TB in unselected adult PLHIV admitted to a district general hospital in Malawi.

The primary outcome is the proportion of people starting TB treatment by the time of death or hospital discharge. The secondary outcomes are all-cause mortality at 56 days from enrolment, proportion of people starting TB treatment within 24 hours from enrolment, and proportion of people with undiagnosed TB. In the CASTLE study we collect a single sputum sample for M. tb culture from participants and undiagnosed TB specifically refers to a person who did not start TB treatment by the time of death or discharge from hospital and has a M. tb cultured from their sputum sample.

Alongside the two trial arms, a third smaller diagnostic cohort arm (1 in 9 of admission days / trial clusters) will explore the range of underlying infectious pathology. The diagnostic cohort does not contribute to trial outcomes.

DETAILED DESCRIPTION:
CASTLE is funded by Wellcome, grant reference 203905/Z/16/Z

ELIGIBILITY:
Inclusion Criteria:

* Requires acute admission to a hospital medical ward at Zomba Central Hospital for any reason
* Is living with HIV (existing or new diagnosis, irrespective of ART status)
* Willing and able to give informed consent

Exclusion Criteria:

* Aged <18 years
* Has been admitted to a medical ward for longer than 18 hours
* Taking TB treatment before admission or has received treatment for TB within the preceding 6 months.
* Has already been in the study during an earlier hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
TB treatment initiation | From time of enrolment into trial to time of discharge from hospital or death (whichever is earlier)
  Proportion of participants started on TB treatment

SECONDARY OUTCOMES:
Mortality | Censored at 56 days from enrolment
  Time (in days) to death from any case.
Undiagnosed TB | From time of enrolment into trial to time of discharge from hospital or death (whichever is earlier)
  Positive sputum culture for mycobacterium tuberculosis at reference lab and participant is not on TB treatment at time of hospital discharge or death.
Same day TB treatment | 24 hours from enrolment
  Proportion of people starting TB treatment within 24 hours of enrollment

OTHER OUTCOMES:
Mortality (measured as a proportion) | 56 days from enrolment
  Proportion of people dying by 56 days from enrolment.
Inpatient mortality | Censored at 56 days for those who are still alive and admitted to hospital at 56 days from enrolment.
  Proportion of people dying prior to hospital discharge
Confirmed TB | From time of enrolment into trial to time of discharge from hospital or death (whichever is earlier)
  The proportion of TB diagnoses that are microbiologically confirmed vs. clinically diagnosed without microbiological confirmation.
Intervention fidelity | 24 hours from enrolment
  Proportion of people randomised to DCXR-CAD plus FujiLAM who have a valid CxR and CAD score recorded, and a FujiLAM result.
Diagnostic accuracy of DCXR-CAD | From time of enrolment into trial to time of discharge from hospital or death (whichever is earlier)
  Sensitivity, specificity, positive and negative predictor value compared to a composite microbiological gold standard.
Prevalence of infectious disease (enhanced diagnostic cohort) | From time of enrolment into trial to time of discharge from hospital or death (whichever is earlier)
  To describe the proportion of patients meeting a clinical or clinical / microbiological description for the following: Sepsis; Invasive bacterial disease; Cryptococcal disease; Pneumocystis jirovecci pneumonia; Bacterial pneumonia; Immune reconstitution inflammatory syndrome (IRIS); HIV treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Rachael M Burke, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Zomba Central Hospital, Zomba, Malawi

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on LSHTM Data Compass.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Burke RM, Nyirenda S, Twabi HH, Nliwasa M, Joekes E, Walker N, Nyirenda R, Gupta-Wright A, Fielding K, MacPherson P, Corbett EL. Design and protocol for a cluster randomised trial of enhanced diagnostics for tuberculosis screening among people living with HIV in hospital in Malawi (CASTLE study). PLoS One. 2022 Jan 10;17(1):e0261877. doi: 10.1371/journal.pone.0261877. eCollection 2022. PMID 35007306

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04545164/SAP_000.pdf